CLINICAL TRIAL: NCT05450003
Title: Effect of Different Irrigation Activating Techniques on Irrigant Penetration Depth Into Root Canals and on Post-Operative Pain After Single-Visit Endodontic Treatment
Brief Title: Effect of Different Irrigation Activating Techniques on Irrigant Penetration Depth and on Post-Operative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Yara Fawzy Kotb Elgazzar, Administrator of endodontics_ faculty of dentistry _Tanta university, Tanta University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: Elgazzar YF1
Record Dates: First submitted 2022-06-18; First posted 2022-07-08 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Irrigation Activation

STUDY DESIGN:
Intervention Model Description: the study will evaluate 3 groups of patients each consists of 10 participants receiving different type of irrigation activation.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- xp endo finisher file (Other)
  Interventions: Device: Irrigation activation using xp endo finisher file , new sonic eddy tip and conventional needle syringe irrigation
- new sonic EDDY system (Other)
  Interventions: Device: Irrigation activation using xp endo finisher file , new sonic eddy tip and conventional needle syringe irrigation
- syringe needle irrigation (Other)
  Interventions: Device: Irrigation activation using xp endo finisher file , new sonic eddy tip and conventional needle syringe irrigation

INTERVENTIONS:
Device: Irrigation activation using xp endo finisher file , new sonic eddy tip and conventional needle syringe irrigation — irrigation activation using 3 different irrigation activation systems including xp endo finisher file , new sonic eddy system and conventional needle syringe irrigation

SUMMARY:
Irrigation activation in endodontics is considered now a very important step for the success of root canal treatment. In this study, the investigator will examine the effect of two recent activation systems ( XP-endo Finisher file and the new sonic EDDY system) in comparison with the conventional needle irrigation on irrigant penetration depth into root canals using radiopaque contrast media and digital radiography and on the postoperative pain after single-visit endodontic treatment using a visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic vital/non vital teeth requiring root canal treatment.
* Teeth with sound periodontal apparatus.
* Teeth without pus or inflammatory exudates draining through the canal.
* Teeth without anatomic variations.
* Teeth with sinus tract.
* Teeth without history of trauma.
* Patients not on analgesics or sedative medication prior to root canal therapy

Exclusion Criteria:

* • Patients with any systemic diseases.

  * Pregnant or lactating patients.
  * Immunocompromised patients.
  * Apparently thin roots in which apical preparation with #40 file would be overzealous.
  * Patient allergic to anything used in this procedure especially rubber dam material and Iohexol (radiographic contrast media).
  * Teeth with calcified canals.
  * Patients with acute apical periodontitis, acute apical abscess, and weeping canals.
  * Necrotic painful teeth with the absence of sinus tract for drainage.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-11-12 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
irrigant penetration depth | through study completion, an average of 3 months
  measurement of irrigant penetration depth using radioaque media and digital radiography
postoperative pain | through study completion, an average of 3 months
  evaluation of postoperative pain using visual analog scale VAS with scores from 0 to 100. score 0 indicated no pain while score 100 indicates maximum pain

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, Egypt

REFERENCES:
- [Derived] Elgazzar YFK, Darrag AM, Attia DAM. Effect of XP-endo Finisher and EDDY activation on post-operative pain after single-visit endodontic treatment: a randomized controlled clinical trial. Sci Rep. 2025 Nov 4;15(1):38476. doi: 10.1038/s41598-025-23628-1. PMID 41188367